CLINICAL TRIAL: NCT01575080
Title: Performance Evaluation of the Contour TS BGMS Using ISO/DIS 15197:2011 Section 8 Study Design and Performance Criteria
Brief Title: Performance Evaluation of Blood Glucose Monitoring System Using ISO Study Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R&D-2011-2012-0.20
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes use Contour TS Blood Glucose Monitoring System.
  Interventions: Device: Contour TS Blood Glucose Monitoring System

INTERVENTIONS:
Device: Contour TS Blood Glucose Monitoring System — Untrained subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick blood and AST of the palm and forearm using the Contour TS Blood Glucose Monitoring System. All BG results are compared to a reference laboratory glucose method.

SUMMARY:
The purpose of this study is to determine if untrained subjects who have diabetes can operate the Blood Glucose Monitoring System (BGMS) and obtain acceptable glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of diabetes
* Be 18 years of age or older
* Be able to speak, read and understand English and understand the Informed Consent document.
* Be willing to complete study procedures

Exclusion Criteria:

* Pregnancy
* Infections or skin disorders at the puncture site (at the discretion of the site professional staff).
* Hemophilia, bleeding disorder, or clotting problems. Persons taking aspirin (81 mg or 325 mg) daily or Plavix® are not reason for exclusion.
* Physical (dexterity), visual, or neurological impairments that would make the person unable to perform testing with the BGM (at the discretion of the site professional staff).
* A condition, in the opinion of the Investigator, would put the subject at risk or influence the conduct of the study or interpretation of the results. The reason for exclusion will be documented by the professional staff.
* Previously participated in a blood glucose monitoring study using Contour TS system or use the Contour TS for personal use when monitoring blood glucose.
* Working for a competitive medical device company or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company
* Working for a medical laboratory, hospital or other clinical setting that involves training on and clinical use of blood glucose monitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 102
Age, Continuous [Median (Full Range); unit: years] | 55 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose Results Within +/- 15mg/dL (<100mg/dL) or Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test fingerstick blood using the Blood Glucose Monitoring System (BGMS). BGMS results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results are used to calculate the number of BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) or +/- 15% (>=100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 102 untrained subjects tested one test strip lot on the Contour TS Blood Glucose Monitoring System.
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 102
Number analyzed (BG test results) | 102
Number of BG Test Results | 84

2. Secondary Outcome: Number of Self-Test Alternative Site (Palm) Blood Glucose Results Within +/- 15mg/dL (<100mg/dL) or Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test Alternative Site (AST) Palm blood using the Blood Glucose Monitoring System (BGMS). BGMS AST palm results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma BG results are used to calculate the number of AST palm BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) or +/- 15% (>=100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 102 untrained subjects tested one test strip lot on the Contour TS Blood Glucose Monitoring System
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 102
Number analyzed (BG test results) | 102
Number of BG Test Results | 78

3. Secondary Outcome: Number of Self-Test Alternative Site (Forearm) Blood Glucose Results Within +/- 15mg/dL (<100mg/dL) or Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-test Alternative Site (AST) Forearm blood using the Blood Glucose Monitoring System (BGMS). BGMS AST forearm results are compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma BG results are used to calculate the number of AST forearm BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) or +/- 15% (>=100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 102 untrained subjects tested one test strip lot using the Contour TS BG Monitoring System. One subject was unable to obtain sufficient sample volume to test. Another subject's meter displayed
Measure: Number; unit: Number of BG Test Results
Units Other Than Participants: BG test results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 102
Number analyzed (BG test results) | 100
Number of BG Test Results | 83

4. Secondary Outcome: Number of Subject Responses That 'Agree' or 'Strongly Agree' With Questionnaire Statements
Description: Subjects will complete short questionnaires to provide feedback on the labeling materials and system ease of use. Subjects may respond 'Strongly Agree' 'Agree' 'Neutral' 'Disagree' 'Strongly Disagree'.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 102
participants
  I found it easy to do a blood test w this meter | 98
  Meter display (test result) is easy to read | 102
  Easy to see and understand the test results | 101
  I like the overall meter design | 80
  Meter is easy to handle | 90
  Easy to handle the individual test strips | 64
  Instructions (User Guide) easy to understand | 97
  Instructions clearly explain how to run a test | 101
  Instructions clearly explain meter error message | 98
  I found this meter easy to use | 100
  I found this meter intuitive | 96
  I found this meter practical | 97

ADVERSE EVENTS:
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 2/102
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=102)
hypoglycemia (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes